CLINICAL TRIAL: NCT01164865
Title: The Subjective Comfort With Multipurpose and Hydrogen Peroxide Lens Care Solutions in Soft Contact Lens Wearers
Brief Title: Subjective Comfort With Multipurpose and Hydrogen Peroxide Lens Care Solutions in Soft Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SMA-09-58
Record Dates: First submitted 2010-07-15; First posted 2010-07-19 (Estimated); Results first posted 2012-10-12 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-09

CONDITIONS: Contact Lens Wear
Keywords: Soft Contact lens; Multi-Purpose Solution; Hydrogen Peroxide
MeSH Terms: interventions — Contact Lenses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- OPTI-FREE RepleniSH (Experimental): OPTI-FREE RepleniSH multipurpose disinfecting solution used with study contact lenses on a daily basis for 2 weeks.
  Interventions: Device: OPTI-FREE RepleniSH multipurpose disinfecting solution; Device: Contact lenses
- Clear Care (Active Comparator): Clear Care contact lens care system used with study contact lenses on a daily basis for 2 weeks.
  Interventions: Device: Clear Care contact lens care system; Device: Contact lenses

INTERVENTIONS:
Device: OPTI-FREE RepleniSH multipurpose disinfecting solution — FDA-approved, multipurpose disinfecting solution used according to provided instructions for cleaning, rinsing, storing, and disinfecting study contact lenses on a daily basis, 2 weeks.
  Other Names: OPTI-FREE® RepleniSH®
  Arms: OPTI-FREE RepleniSH
Device: Clear Care contact lens care system — FDA-approved, hydrogen peroxide-based, lens care system used according to provided instructions for cleaning, disinfecting, daily protein removing, and storage of study contact lenses on a daily basis, 2 weeks.
  Other Names: Clear Care®
  Arms: Clear Care
Device: Contact lenses — Contact lenses per subject's habitual brand and prescription worn every day for the duration of the study, 14 days, on a daily wear basis without scheduled replacement.

SUMMARY:
The purpose of this study was to assess comfort in soft contact lens wearers.

ELIGIBILITY:
Inclusion Criteria:

* Wear silicone hydrogel contact lenses on a daily wear basis;
* Currently using OPTI-FREE RepleniSH contact lens solution;
* Report comfort above 75 on a Visual Analog Scale at the Baseline Visit;
* Read, sign, and date IRB-approved informed consent and the privacy document;
* Be generally healthy and have normal ocular health;
* Be be willing to follow the study procedures and visit schedule;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Use of additional lens cleaners;
* Known sensitivity to any ingredient in either of the test articles;
* Systemic or ocular disease or disorder (except refractive error) that would negatively affect the conduct or outcome of the study;
* Prior (within 7 days of enrollment) or current ocular infections;
* Clinically significant lash or lid abnormality;
* History of ocular surgery/trauma within the last 6 months;
* Use of any topical ocular or systemic antibiotics or corticosteroids within 7 days of enrollment;
* Participation in any other ophthalmic drug or device clinical trial within 30 days of enrollment;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from two US study centers.
Period: Overall Study
Arm/Group | OPTI-FREE RepleniSH | Clear Care
Started | 39 | 39
Completed | 37 | 38
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OPTI-FREE RepleniSH | Clear Care | Total
Number analyzed (Participants) | 39 | 39 | 78
Age Continuous [Mean (Standard Deviation); unit: years] | 37.1 (12.27) | 41.5 (9.59) | 39.3 (11.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 26 | 55
  Male | 10 | 13 | 23
Region of Enrollment [Number; unit: participants]
  United States | 39 | 39 | 78

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Ocular Comfort Rating at 2 Weeks
Description: Ocular comfort was rated by the participant on a continuous visual analog scale from 0-100, where 0=extremely uncomfortable, 50=neither comfortable nor uncomfortable, and 100=extremely comfortable. The participant marked a horizontal line across the scale at the point that best described "how your eyes feel right now."
Time Frame: Baseline (Day 0), 2 weeks
Population: All participants who received regimen, satisfied the inclusion/exclusion criteria, and completed the 14-day treatment period, including completion of the Visit 2 evaluations.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | OPTI-FREE RepleniSH | Clear Care
Number analyzed (Participants) | 37 | 38
Units on a scale | -8.20 [-13.84 to -2.55] | -7.14 [-12.74 to -1.54]

2. Primary Outcome: Likert Questionnaire Scores at 2 Weeks
Description: The Likert Questionnaire included 8 questions on selected comfort measures. All responses were recorded on a 5-point scale, where 1=Strongly Disagree, 2=Disagree, 3=Undecided, 4=Agree, and 5=Strongly Agree.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | OPTI-FREE RepleniSH | Clear Care
Number analyzed (Participants) | 37 | 38
Units on a scale
  I can comfortably wear my lenses | 4.20 [3.96 to 4.44] | 4.24 [4.00 to 4.48]
  My lenses stay moist from morning to evening | 3.60 [3.28 to 3.92] | 3.69 [3.37 to 4.01]
  The solution I use feels gentle on my eyes | 4.00 [3.75 to 4.25] | 3.66 [3.41 to 3.91]
  My lenses feel fresh | 3.79 [3.52 to 4.05] | 4.03 [3.77 to 4.29]
  At the end of the day, my vision is clear | 3.54 [3.20 to 3.88] | 3.86 [3.52 to 4.19]
  When I put my lenses in, they feel comfortable | 4.05 [3.78 to 4.33] | 4.03 [3.76 to 4.30]
  I like the way this product feels during handling | 4.09 [3.84 to 4.34] | 3.66 [3.42 to 3.91]
  My lenses feel moist | 3.84 [3.56 to 4.12] | 3.64 [3.36 to 3.92]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study: 5 months, 3 weeks.
Description: The safety population included all enrolled and exposed participants.
Arm/Group | OPTI-FREE RepleniSH | Clear Care
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 0/39 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Alcon reserves the right of prior review of any publication or presentation of information related to the study.